CLINICAL TRIAL: NCT01989702
Title: The Effect of a Probiotic-based Product on Blood Pressure and Other Known Risk Factors Linked to Cardiovascular Diseases.
Brief Title: Effect of a Probiotic-based Product on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ProMeta
Record Dates: First submitted 2013-11-07; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Fermented blueberry product (Active Comparator)
  Interventions: Other: Fermented blueberry drink; Other: Sachets with placebo powder
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo drink; Other: Sachets with placebo powder
- Probiotic bacteria (Active Comparator)
  Interventions: Other: Placebo drink; Other: Sachets with probiotic bacterial powder

INTERVENTIONS:
Other: Fermented blueberry drink
  Arms: Fermented blueberry product
Other: Placebo drink
  Arms: Placebo; Probiotic bacteria
Other: Sachets with probiotic bacterial powder
  Arms: Probiotic bacteria
Other: Sachets with placebo powder
  Arms: Fermented blueberry product; Placebo

SUMMARY:
The aim of the present study was to examine the efficacy of a probiotic-based product on either reducing hypertension or preventing a high normal blood pressure from reaching hypertensive levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals at the age of 40-75 years.
* Blood-pressure >140/90 mmHg that has been confirmed at 2-3 separate occasions or represents the mean value of a 24-hour measurement.
* Triglycerides >1,7 mmol/L and/or HDL <1 mmol/L (men)/1,29 mmol/L (women).
* Fasting plasma glucose levels >5,6 mmol/L and/or waist circumference >102 cm (men)/88 cm (women).
* BMI <40.

Exclusion Criteria:

* Medically treated allergy or allergy to any of the ingredients of the study product.
* Medication for high levels of blood lipids.
* Metabolic disease, such as type one diabetes.
* Confirmed diseases of the heart, liver of kidneys.
* Chronic inflammatory disease requiring medication.
* Pregnant or nursing.
* Regular intake of other probiotic products (5-7 days per week during the last three months before inclusion into the study).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in systolic and diastolic blood pressure after 3 months of probiotic intervention | Baseline, 3 months

SECONDARY OUTCOMES:
Changes from baseline of blood parameters, such as inflammatory markers and blood lipids, linked to increased risk for cardiovascular diseases | Baseline, 3 months

OTHER OUTCOMES:
Effect of study product on intestinal microbiota as analysed in fecal samples | Baseline, 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Malmo, Sweden